CLINICAL TRIAL: NCT02742233
Title: A Controlled Clinical Trial of Dipeptidyl Peptidase 4 Inhibition Facilitate Healing of Diabetic Ulcers
Brief Title: Dipeptidyl Peptidase 4 Inhibition Facilitate Healing of Diabetic Ulcers
Acronym: DPP4i
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Long Min,MD (Other)
Responsible Party: Sponsor-Investigator, Long Min,MD, Principal Investigator, Xinqiao Hospital of Chongqing
Organization: Xinqiao Hospital of Chongqing (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XinqiaoH
Record Dates: First submitted 2016-03-24; First posted 2016-04-18 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-01

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; Wound Healing; Dipeptidyl Peptidase 4 Inhibition
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- saxagliptin (Experimental): saxagliptin & Regular treatment:
  saxagliptin, brand name，Bristol-Myers, Squibb, dose: 5mg, po, qd
  Interventions: Drug: saxagliptin
- placebo (Placebo Comparator): placebo & Regular treatment:
  placebo, dose: 5mg, po, qd
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: saxagliptin — Qualifying Period: Participants will receive regular treatment for diabetic ulcer without DPP4i.
  Treatment Period: Participants will receive saxagliptin with regular treatment
  Other Names: ONGLYZA
  Arms: saxagliptin
Drug: placebo — Qualifying Period: Participants will receive regular treatment for diabetic ulcer without DPP4i.
  Treatment Period: Participants will receive placebo with regular treatment
  Other Names: dummy pills
  Arms: placebo

SUMMARY:
To investigate the effect of Dipeptidyl Peptidase 4 Inhibition on wound healing in patients with diabetic foot ulcers, the investigators randomly divided the participants into two groups: saxagliptin with regular treatment group，placebo with regular treatment group. The clinical data are collected at the given time point. This study aimed to observe the potential protective effect of DPP4i on diabetic ulcers.

DETAILED DESCRIPTION:
Groups:

Diabetic ulcers, saxagliptin + Regular treatment.

Diabetic ulcers, placebo + Regular treatment.

Time Point:

Initial treatment;

Post-treatment ( 1w );

Post-treatment ( 2w );

Post-treatment ( 4w );

Completely healed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus according to World Health Organization criteria ( treatment with insulin or an oral hypoglycemic agent, twice random glucose measurements major than 200 mg/dl, or a fasting glucose major than 140 mg/dl)
* Ulcer located on the legs or feet, stage III or IV (Wagner Classification System)
* The subject agrees to comply with study protocol requirements and all follow up visit requirements.

Exclusion Criteria:

* Uncontrolled diabetes
* Ulcer infection
* Non-diabetic ulcers Orthopedic or neuromuscular pathologic conditions

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Completely healing time of the participants'target ulcer during the treatment period. | 16 weeks
  Complete ulcer closure is defined as 100% skin re-epithelialization

SECONDARY OUTCOMES:
Proportion of participants with complete healing during the treatment period. | 16 weeks
  Complete ulcer closure is defined as 100% skin re-epithelialization

OTHER OUTCOMES:
Net change from baseline in laboratory test results | Baseline, weeks 1, 2,4,
New ulcers | 16 weeks
  new ulcers among the participants during treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Hongting Zheng, Ph.D, Principal Investigator — Department of Endocrinology,The Second Affiliated Hospital, Third Military Medical University, Chongqing, People's Republic of China.
Locations (1):
- The Second Affiliated Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
age，the grade of the diabetic ulcers, sex, diabetes duration, healing time, treatment. ect